CLINICAL TRIAL: NCT05375903
Title: A Phase 1, Open-label, Dose-escalation Study to Investigate the Safety, Tolerability, and Pharmacokinetics of UGN-301 (Zalifrelimab) Administered Intravesically as Monotherapy and in Combination With Other Agents in Patients With Recurrent NMIBC
Brief Title: A Phase 1 Dose-escalation Study of UGN-301 in Patients With Recurrent Non-muscle Invasive Bladder Cancer (NMIBC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UroGen Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UR001
Record Dates: First submitted 2022-05-05; First posted 2022-05-17 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Non-muscle Invasive Bladder Cancer; NMIBC; Carcinoma in Situ of Bladder; Bladder Cancer; Urothelial Carcinoma Bladder; Urothelial Carcinoma Recurrent
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Urinary Bladder Neoplasms | interventions — Imiquimod; Gemcitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- UGN-301 monotherapy dose escalation (Arm A) (Experimental): Dose escalation of UGN-301 monotherapy in patients with recurrent NMIBC with high grade (HG) Ta and/or T1 disease and/or CIS or recurrent intermediate risk (IR) low grade (LG) Ta and/or T1 disease.
  Interventions: Drug: UGN-301
- UGN-301 dose escalation + UGN-201 combination (Arm B) (Experimental): Dose escalation of UGN-301 in combination with a fixed dose of UGN-201 in patients with recurrent NMIBC with HG Ta and/or T1 disease and/or CIS.
  Interventions: Drug: UGN-301; Drug: UGN-201
- UGN-301 dose escalation + gemcitabine combination (Arm C) (Experimental): Dose escalation of UGN-301 in combination with a fixed dose of gemcitabine in patients with recurrent NMIBC with HG Ta and/or T1 disease and/or CIS.
  Interventions: Drug: UGN-301; Drug: Gemcitabine

INTERVENTIONS:
Drug: UGN-301 — Induction Period: Intravesical administration once weekly for 6 weeks.
  Optional Maintenance Period: Intravesical administration once every 3 months (at 6, 9, and 12 months after the start of treatment).
  Other Names: UGN-301 (zalifrelimab) intravesical solution
Drug: UGN-201 — Induction Period: Intravesical administration once weekly for 6 weeks.
  Optional Maintenance Period: Intravesical administration once every 3 months (at 6, 9, and 12 months after the start of treatment).
  Other Names: UGN-201 (imiquimod) intravesical solution
  Arms: UGN-301 dose escalation + UGN-201 combination (Arm B)
Drug: Gemcitabine — Induction Period: Intravesical administration once weekly for 6 weeks.
  Optional Maintenance Period: Intravesical administration once every 3 months (at 6, 9, and 12 months after the start of treatment).
  Arms: UGN-301 dose escalation + gemcitabine combination (Arm C)

SUMMARY:
This study is being conducted to evaluate the safety and determine the recommended Phase 2 dose (RP2D) of UGN-301 (zalifrelimab) administered intravesically as monotherapy and in combination with other agents in patients with recurrent NMIBC.

DETAILED DESCRIPTION:
This master protocol will comprise multiple treatment arms designed to independently investigate intravesical delivery of UGN-301 either as monotherapy or in combination with other agents. Initial study treatment arms will include:

* UGN-301 monotherapy
* UGN-301 + UGN-201 (imiquimod) in combination
* UGN-301 + gemcitabine in combination

Additional study treatment arms investigating UGN-301 in combination with other agents may be added in the future.

The study will evaluate escalating doses of UGN-301 to determine the biologically effective dose (BED) and maximum tolerated dose (MTD) of UGN-301 either as monotherapy or in combination with other agents.

When evaluated in combination with other agents, the UGN-301 dose will begin at least 1 dose level lower than the highest dose level cleared in the monotherapy arm, or 1 dose level lower than the RP2D.

Eligible patients in each study treatment arm will enter a 12-week Induction Period.

Patients with noninvasive papillary carcinoma and/or tumor that invades the lamina propria (Ta and/or T1) who do not have disease recurrence and patients with carcinoma in situ (CIS) who have a complete response (CR) at 3 months after the start of treatment will return to the clinic for a Safety Follow-up Visit at 6 months after the start of treatment.

Ta/T1 patients without disease recurrence and CIS patients with CR at 6 months may enter an Optional Maintenance Period of up to 9 months.

ELIGIBILITY:
Inclusion Criteria:

1. Able to give informed consent.
2. Arm A: Have confirmed recurrent NMIBC with HG Ta and/or T1 disease and/or CIS or recurrent IR LG Ta and/or T1 disease.

   Arm B: Have confirmed recurrent NMIBC with HG Ta and/or T1 disease and/or CIS. Arm C: Have confirmed recurrent NMIBC with HG Ta and/or T1 disease and/or CIS.
3. Patients with HG Ta and/or T1 disease and/or CIS must meet one of the following criteria:

   • Have Bacillus Calmette-Guérin (BCG)-unresponsive disease, defined as 1) persistent or recurrent CIS alone or with recurrent Ta/T1 disease within 12 months of completion of adequate BCG therapy, or 2) recurrent HG Ta/T1 disease within 6 months of completion of adequate BCG therapy, or 3) HG T1 disease at the first evaluation following a BCG induction course.

   Notes: Adequate BCG therapy is defined as at least 5 of 6 doses of an initial induction course plus 1) at least 2 of 3 doses of maintenance therapy or 2) at least 2 of 6 doses of a second induction course. Patients with BCG-unresponsive disease also must be unwilling or unfit to undergo radical cystectomy.
   * Have otherwise failed adequate BCG therapy (eg, recurrence > 6 months [papillary] or > 12 months [CIS] after last BCG exposure).
   * Are BCG intolerant, defined as the inability to tolerate at least one full induction course of BCG.
   * Have HG Ta disease with tumors ≤ 3 cm and failed at least one previous course of therapy (eg, adjuvant intravesical chemotherapy).
4. Have all papillary tumors visible by white light resected, and obvious areas of CIS fulgurated during Screening or within 6 weeks before Screening. Note: Blue light cystoscopy is not permitted.
5. Eastern Cooperative Oncology Group (ECOG) status ≤ 2.
6. Absence of concomitant upper tract urothelial carcinoma (UTUC) or urothelial carcinoma (UC) within the prostatic urethra. Freedom from upper tract disease (if clinically indicated) as indicated by no evidence of upper tract tumor by either intravenous pyelogram, retrograde pyelogram, computerized tomography (CT) urogram with or without contrast, or magnetic resonance imaging (MRI) urogram with or without contrast performed within 6 months of enrollment.
7. Patients with prostate cancer on active surveillance at very low, low, or intermediate risk for progression, defined as Gleason Grade Group 1 or 2, Gleason score ≤ 7, with prostate-specific antigen < 20 ng/dL, and cT1-cT2b (NCCN, 2023) are permitted to be in the study at the discretion of the investigator (see exclusion criterion 8).
8. Female patients of childbearing potential must use maximally effective birth control during the period of therapy, must be willing to use contraception for 1 month following the last administration of study drug and must have a negative urine or serum pregnancy test upon entry into this study. Otherwise, female patients must be postmenopausal (no menstrual period for a minimum of 12 months) or surgically sterile. "Maximally effective birth control" means that the patient, if sexually active, should be using a combination of 2 methods of birth control that are approved and recognized to be effective by health authorities.
9. Male patients must be surgically sterile or willing to use 2 highly effective forms of birth control upon enrollment, during the course of the study, and for 1 month following the last study drug instillation.
10. Has adequate organ and bone marrow function within 14 days of treatment initiation as determined by routine laboratory tests outlined below:

    * Leukocytes ≥ 3,000/μL;
    * Absolute neutrophil count (ANC) ≥ 1,500/μL;
    * Platelets ≥ 100,000/μL;
    * Hemoglobin ≥ 9.0 g/dL;
    * Total bilirubin ≤ 1.5 × upper limit of normal (ULN);
    * Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 2.5 × ULN;
    * Alkaline phosphatase (ALP) ≤ 2.5 × ULN;
    * Estimated creatinine clearance ≥ 30 mL/min calculated using the Cockcroft-Gault equation.
11. Has a life expectancy > 12 months.

Exclusion Criteria:

1. Current or previous evidence of muscle invasive, locally advanced nonresectable, or metastatic urothelial carcinoma (ie, T2, T3, T4 and/or stage IV).
2. Current systemic therapy for bladder cancer.
3. Prior therapy with an anti-cytotoxic T lymphocyte antigen 4 (CTLA-4), anti-programmed cell death 1 (PD-1), anti-PD-ligand 1 (L1) agent, or with an agent directed to another co-inhibitory T-cell receptor.
4. Active infection requiring systemic therapy including urinary tract infection (once satisfactorily treated, patients can enter the study).
5. Active systemic autoimmune disease that required systemic treatment in the past 2 years. Short courses of steroids (≤ 14 days) for medical reasons without anticancer intent (eg, atopic dermatitis, psoriasis, infection, allergic reaction) are permitted if the last dose was ≥ 4 weeks before the first dose of study treatment.
6. Women who are pregnant or nursing.
7. Any medical psychological, familial, sociological, or geographical condition that, in the opinion of the Investigator, would preclude participation in the study.
8. History of malignancy of other organ system within the past 5 years, except previously treated UTUC, basal cell carcinoma or squamous cell carcinoma of the skin, and/or prostate cancer under active surveillance (see inclusion criterion 8).
9. Patients who cannot tolerate intravesical dosing or intravesical surgical manipulation.
10. Intravesical therapy within 4 weeks before starting study treatment.
11. Has participated in a study of an investigational agent and received study therapy or received investigational device within 4 weeks before the first dose of study treatment.
12. Has received an immune modulator therapy within 5 half-lives of starting study treatment.
13. Has received a vaccine within 2 weeks before starting study treatment.
14. Has a known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2026-01-09 (Actual); Study Completion 2026-01-09 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs) and treatment-emergent adverse events (TEAEs) | Up to 15 months
  The number of patients with each type of event will be summarized.
Concentration of UGN-301 in blood and urine | 6 weeks
  Data will be summarized using descriptive statistics.
Complete response rate (CRR) | 3 months
  CRR is defined as the proportion of CIS patients who achieved CR at the Week 12 (3-month) Visit.
Recurrence-free survival (RFS) rate | 3 months
  RFS rate is defined as the proportion of patients with Ta/T1 disease who are recurrence-free at the Week 12 (3-month) Visit.

SECONDARY OUTCOMES:
Presence of anti-drug antibodies (ADA) in serum | 3 months
  The number of patients with ADA will be summarized.
UGN-301 maximum serum concentration (Cmax) following single and repeat dose administration | 6 weeks
  Data will be summarized using descriptive statistics.
UGN-301 area under the concentration-time curve (AUC) following single and repeat dose administration | 6 weeks
  Data will be summarized using descriptive statistics.
UGN-301 time to maximum serum concentration (tmax) following single and repeat dose administration | 6 weeks
  Data will be summarized using descriptive statistics.
UGN-301 terminal half-life (t1/2) following single and repeat dose administration | 6 weeks
  Data will be summarized using descriptive statistics.
UGN-301 concentration in serum at the end of a dosing interval (Ctau) following single and repeat dose administration | 6 weeks
  Data will be summarized using descriptive statistics.
Concentration of UGN-201 and its metabolites in blood and urine | 6 weeks
  Data will be summarized using descriptive statistics.
UGN-201 Cmax following single and repeat dose administration | 6 weeks
  Data will be summarized using descriptive statistics.
UGN-201 AUC following single and repeat dose administration | 6 weeks
  Data will be summarized using descriptive statistics.
UGN-201 tmax following single and repeat dose administration | 6 weeks
  Data will be summarized using descriptive statistics.
UGN-201 t1/2 following single and repeat dose administration | 6 weeks
  Data will be summarized using descriptive statistics.
UGN-201 Ctau following single and repeat dose administration | 6 weeks
  Data will be summarized using descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Mirkin, MD, Study Director — UroGen Pharma
Locations (13):
- United States (7):
  - Arkansas Urology, Little Rock, Arkansas
  - UCLA - University of California, Los Angeles, California
  - Florida Urology Partners, LLC, Tampa, Florida
  - Johns Hopkins University, Baltimore, Maryland
  - Manhattan Medical Research, New York, New York
  - Clinical Research Solutions, Middleburg Heights, Ohio
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
- Italy (3):
  - I.R.C.C.S. Ospedale San Raffaele, Milan
  - National Tumor Institute Fondazione G. Pascale, Naples
  - Istituto Oncologico Veneto, Padua
- Spain (3):
  - NEXT Oncology IOB- Hospital Quironsalud Barcelona, Barcelona
  - Hospital Clinic de Barcelona Instituto Clinic de Nefrologia y Urologia (ICNU), Barcelona
  - NEXT Oncology- Hospital Quironsalud Mardrid, Madrid